CLINICAL TRIAL: NCT03232476
Title: Effect of Mechanical Loading With PTH on Cortical Bone
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unsuccessful recruitment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joy Tsai, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P001094
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Loaded upper extremity (Other): This is a one-arm study. In postmenopausal women prescribed teriparatide for osteoporosis treatment, enrolled subjects will perform voluntary loading exercises on one upper extremity. A data logger device will assist in recording exercises and determining goal force during the exercises. Each subject's non-loaded upper extremity will serve as a control.
  Interventions: Device: Upper extremity voluntary loading

INTERVENTIONS:
Device: Upper extremity voluntary loading — Subjects who are prescribed teriparatide by their healthcare provider may enroll in this study. The study intervention consists of loading one upper extremity. Subjects will be trained on how to perform the upper extremity exercises at home. Subjects will be expected to perform the exercises 3 days per week using one arm, with each session consisting of 100 loading cycles lasting a total of approximately 2 minutes each day.

SUMMARY:
Clinical trial to investigate effect of voluntary upper extremity loading in combination with anabolic osteoporosis therapy.

ELIGIBILITY:
Inclusion Criteria:

* women aged 45+
* postmenopausal
* osteoporotic with high risk of fracture

Exclusion Criteria:

* no significant previous use of bone health modifying treatments

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
radius bone mineral density | 12 month change

CONTACTS AND LOCATIONS:
Overall Officials: Joy Tsai, MD, Principal Investigator — MGH